CLINICAL TRIAL: NCT06766032
Title: Comparison of the Performance and Effectiveness of Two Transfusion-Saving Devices: Cell-Saver for Red Blood Cell Reinfusion and SAME for Red Blood Cell and Platelet Reinfusion
Brief Title: Comparison of the Performance and Effectiveness of Two Transfusion-Saving Devices: Cell-Saver and SAME
Acronym: SAME-CELL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AR_2024_001
Record Dates: First submitted 2024-12-16; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Surgery Under Extra Corporeal Circulation; Cardiac Surgery Requiring Cardiopulmonary Bypass
Keywords: cell-saver; auto-transfusion; platelet transfusion; blood saving techniques
MeSH Terms: interventions — Operative Blood Salvage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cell-Saver group: Patients for whom the Cell-saver device is used during cardiac surgery.
  Interventions: Device: CELL-Saver
- SAME group: Patients for whom the SAME device is used during cardiac surgery.
  Interventions: Device: SAME

INTERVENTIONS:
Device: CELL-Saver — The Cell-saver device allows for red blood cell reinfusion during cardiac surgery.
  Groups: Cell-Saver group
Device: SAME — The SAME device allows for red blood cell and platelet reinfusion during cardiac surgery.
  Groups: SAME group

SUMMARY:
An observational study comparing two systems of perioperative blood recovery in cardiac surgery, one system allowing red blood cell reinfusion and one system allowing red blood cell and platelet reinfusion. The objective is to evaluate whether platelet recovery provides better quality of hemostasis during and after surgery, improving transfusion savings, and whether it reduces postoperative complications and the length of stay in the intensive care unit and in the hospital.

DETAILED DESCRIPTION:
° Primary outcome of the study : The primary outcome of the study is to compare the evolution of perioperative platelet count based on the type of blood recovery used, either SAME or Cell-Saver.

The main outcome measure is the difference between the preoperative and immediate postoperative platelet counts (delta platelet) for each patient between the SAME and Cell-Saver groups.

° Secondary outcomes of the study:

The secondary outcomes are to evaluate, from the preoperative period until day 28 postoperatively:

* The post-operative platelet count between days 1 and 5
* The frequency of perioperative and postoperative transfusions, including the number and type of blood products transfused
* The use of derivative medications (fibrinogen, prothrombin complex concentrates)
* The volume of postoperative bleeding
* The frequency of postoperative events (infectious, renal, thromboembolic, hemorrhagic)
* The length of stay in the intensive care unit and in the hospital
* The frequency of treatment for postoperative anemia with iron or erythropoiesis-stimulating agents.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled cardiac surgery under cardiopulmonary bypass with a predicted duration of more than 2 hours, or surgery of the aortic arch, redo surgery, multiple aorto-coronary bypasses (>2), or combined surgery (valvular and coronary).

Exclusion Criteria:

* Pre-existing constitutional or acquired bleeding disorder (hemophilia A or B, von Willebrand disease, myelodysplastic/myeloproliferative syndrome)
* Patients with sepsis, a malignant tumor at the surgical site, or contamination of recovered blood with biological fluids/antiseptics/distilled water/local antibiotics/hemostatic agents.
* Organ transplantation and planned circulatory support in the preoperative period
* Uni-bi-ventricular artificial heart
* Reoperation in a patient already included in the study
* Patient refusing blood transfusion
* Pregnant women
* Legally Protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated by the cardiac surgery department of Nantes University Hospital who undergo a cardiovascular procedure with cardiopulmonary bypass considered to be at high risk for bleeding; (prolonged cardiopulmonary bypass >2 hours, aortic arch surgery, history of redo cardiac surgery, combined surgery, multiple portocoronary bypasses). Procedures for which a perioperative blood recovery device (SAME or Cell-Saver) has been used, with the choice of the blood recovery technique at the discretion of the medical team.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Difference between the preoperative and immediate postoperative platelet counts (delta of platelet) for each patient | up to 1 week
  The main outcome measure is the difference between the preoperative and immediate postoperative platelet counts (delta platelet) for each patient in the Cell-saver group or in the SAME group.

SECONDARY OUTCOMES:
Postoperative platelet | 5 days
  Postoperative platelet count between day 1 and day 5
Perioperative and postoperative transfusions | 28 days
  Frequency of perioperative and postoperative transfusions, number and type of blood products transfused from surgery (day 1) to 28 days after surgery
Derivative medications | 28 days
  Use of derivative medications (fibrinogen, prothrombin complex concentrates) from surgery (day 1) to 28 days after surgery
Postoperative bleeding | 28 days
  Volume of postoperative bleeding from surgery (day 1) to 28 days after surgery
Postoperative events | 28 days
  Frequency of postoperative events (infectious, renal, thromboembolic, hemorrhagic) from surgery (day 1) to 28 days after surgery
Durations of stays | 28 days
  Duration of stays in the intensive care unit and in the hospital from surgery (day 1) to 28 days after surgery
Postoperative anemia | 28 days
  Frequency of treatment for postoperative anemia with iron or erythropoiesis-stimulating agents from surgery (day 1) to 28 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mickaël Vourc'h, MD-PhD, Principal Investigator — Nantes HU
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided